CLINICAL TRIAL: NCT03252678
Title: Efficacy of Self-education Program for Advanced Care Planning: A Randomized Controlled Trial
Brief Title: Efficacy of Self-education Program for Advanced Care Planning(RCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Institute of Health, Korea (Other Government); National Clinical Research Coordination Center, Seoul, Korea (Other Government); Ewha Womans University Mokdong Hospital (Other); Ulsan University Hospital (Other); Keimyung University Dongsan Medical Center (Other); Asan Medical Center (Other); Gangneung Asan Hospital (Other); Korea University Anam Hospital (Other); Daegu Fatima Hospital (Other); National Evidence-Based Healthcare Collaborating Agency (Other Government); Pohang Semyeong Christianity Hospital (Unknown)
Responsible Party: Principal Investigator, Young Ho Yun, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HC15C1391-3
Record Dates: First submitted 2017-07-13; First posted 2017-08-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Advanced Cancer
Keywords: Advanced Care Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Book and Videos about ACP (Experimental): Subjects in experimental group get a book of 45 pages and three videos about advanced care planning based on Smart Management Strategy for Health (SMASH). After they finish reading and watching the materials, they fill out the questionnaire.
  Interventions: Other: a book and videos about ACP
- A Book and Videos about Pain Control (Active Comparator): Subjects in the group get a book and two videos about pain control for cancer patients. After they finish reading and watching the materials, they fill out the questionnaire.
  Interventions: Other: a book and videos about pain control

INTERVENTIONS:
Other: a book and videos about ACP — A book and three videos about advanced care planning are provided for self-education
  Arms: A Book and Videos about ACP
Other: a book and videos about pain control — A book and three videos about pain control for cancer patients are provided for self-education
  Arms: A Book and Videos about Pain Control

SUMMARY:
This study verifies efficacy of Self-education program for advanced care planning. Half of participants will receive a book and videos about advanced care planning while the other half will receive a book and videos about pain control for cancer patients.

DETAILED DESCRIPTION:
This study validates effectiveness of educational materials that the investigators developed due to the rates of completing advanced care planning are considerably low and patients relatively less less preferred to receive palliative care and hospice at terminal status, which is led by the lack of information available to patients; whether these decision aids change end-of-life care preference, elevate the preference of patients toward advanced care planning, reduce the burden of decision making compare to educational resources that are currently available.

Previous studies inform that educational video about advanced care planning increases the knowledge of care for life prolongation, and affects the preference towards care for life prolongation and palliative care. However, being no resources are provided and orally explained, patients in the control group don't have enough time to fully aware of the information, also, since those studies are done mostly in the western countries, 'discussing with family members or guardians' part is missing, which is critical under contemporary Korean medical society. This study provides educational resources to both the intervention group and the control group and identifies if advanced care planning is discussed with family members or guardians.

Primary outcome of this study is end-of-life care preference. Participants of this study will fill out the baseline questionnaire about end-of-life care preference, end-of-life discussion and documentation, knowledge of ACP, etc. After that, participants will be allocated equally into the intervention group and the control group. The intervention group will receive a book and videos about advanced care planning which are based on Smart Management Strategy for Health(SMASH). The control group will receive a book and videos about pain control for cancer patients that were provided by Korea National Cancer Center. After reading and watching the educational materials, patients will get another questionnaire about knowledge of ACP, satisfaction on the materials, end-of-life care preference, and decision role preference. Participants will read and watch the materials for about 6-8 weeks and then they will be asked to complete another questionnaire which includes every questions from the baseline and post-intervention. The result from all three questionnaires (baseline, post-intervention, 7-week questionnaire) will be compiled and be compared with one another.

ELIGIBILITY:
Inclusion Criteria:

* Subject 20 years old and more
* Subject who understands the purpose of the study and signs with informed consent form
* Subject with advanced cancer
* Subject who knows he/she is diagnosed with advanced cancer

Exclusion Criteria:

* Inability to speak, understand, or write Korean
* Inability to understand the contents of the provided materials due to poor eyesight and hearing
* Medical conditions that would limit adherence to participation of the clinical trial (as confirmed by their referring physician; e.g. dyspnea, depression and other mental disorders)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in End-of-life Care Preference | Baseline, within 1 week, 7 weeks
  Comparison the result of End-of-life Care Preference questionnaire

SECONDARY OUTCOMES:
Changes in Hospital Anxiety and Depression Scale | Baseline, 7 weeks
  Comparison the result of Hospital Anxiety and Depression Scale
Changes in Decision Conflict | Baseline, 7 weeks
  Comparison the result of decision conflict questionnaire
Changes in EOL care Discussion and Documentation | Baseline, 7 weeks
  Comparison the result of EOL care Discussion and Documentation questionnaire
Changes in Satisfaction on educational materials | Baseline, 7 weeks
  Comparison Satisfaction on educational materials questionnaire
Changes in Decisional Role Preference | Baseline, 7 weeks
  Comparison the result of decisional role preference questionnaire
Changes in Knowledge of CPR | Baseline, 7 weeks
  Comparison the result of knowledge of CPR questionnaire
Intention to document advance care planning | Baseline, 7 weeks
  Comparison the result of advance care planning questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Young Ho Yun, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University, Seoul, South Korea